CLINICAL TRIAL: NCT04965142
Title: Feasibility of a Home-Based Exercise Program in Lung and Liver Transplant Recipients for Management of Post-Transplant Metabolic Syndrome: a Pilot Randomized Controlled Trial
Brief Title: Feasibility of a Home Exercise Program to Manage Post-transplant Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian National Transplant Research Program (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-5185
Record Dates: First submitted 2021-06-17; First posted 2021-07-16 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Metabolic Syndrome
Keywords: Lung Transplant Recipients; Liver Transplant Recipients; Exercise Training
MeSH Terms: conditions — Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Lung and liver transplant recipients will be randomized to home exercise group versus usual care group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home Exercise Group (Experimental): The home-based exercise group will be asked to exercise 3 to 5 times per week (≥ 150 minutes of aerobic exercises (i.e. walking, cycling, or treadmill) of at least moderate intensity) and to also complete resistance training (resistance bands or free weights) at least twice weekly over a 12-week period supervised by an exercise professional. The resistance training will be personalized, aiming for 6 to 10 exercises targeting the major muscle groups, progressing to 3 sets of 8 to 12 repetitions. Exercise prescriptions will be developed and monitored by an exercise professional with weekly follow-up meetings and supported with a web application (Physiotec) that allows customizable exercise prescriptions, tracking of exercise completion, and video tutorials. Participants will receive one counselling session on healthy eating and physical activity at the start of the study along with an exercise manual.
  Interventions: Behavioral: Exercise Training
- Control Group (No Intervention): Participants will receive one counselling session on healthy eating and physical activity at the start of the study.

INTERVENTIONS:
Behavioral: Exercise Training — The intervention group will be asked to complete aerobic exercises 3 to 5 times per week (≥ 150 minutes of at least moderate aerobic intensity) and resistance training at least twice a week over a 12-week period.
  Arms: Home Exercise Group

SUMMARY:
Post-transplant metabolic syndrome (PTMS) affects about 50% liver transplant (OLT) and 25% lung transplant (LTx) recipients at 12-18 months post-transplant. PTMS (comprised of glucose intolerance, obesity, hypercholesterolemia and hypertension) has been associated with increased risk for cardiovascular morbidity and long-term survival. Exercise studies in the early post-transplant period have shown some benefits on PTMS risk factors with facility-based training, but it remains unclear if exercise can be sustained in the home environment with sufficient adherence or training intensity to impact PTMS beyond the early post-transplant period. Objectives: 1) To evaluate the feasibility of a three-month individualized, virtual home-based exercise training program in OLT and LTx recipients starting at 1 year post-transplant. 2) To assess estimates of intervention efficacy on elements of PTMS, insulin resistance, exercise self-efficacy, and health related quality of life (HRQL). Methods: 20 OLT and 20 LTx recipients with 2 or more PTMS risk factors at 12-18 months post-transplant will be randomized to a home-based exercise program versus usual care. The exercise group will undergo aerobic training 3 to 5 times per week with resistance training at least twice weekly over a 12-week period. Exercises will be demonstrated by a qualified exercise professional during the first visit with weekly phone and video calls to guide exercise progression, ease communication and promote exercise self-efficacy and adherence based on guiding behavioral principles. As secondary measures, PTMS, insulin resistance, body composition (optional), HRQL, and assessment of self-efficacy will be assessed at baseline and 12-weeks.

DETAILED DESCRIPTION:
Both LTx and OLT recipients have several common risk factors for PTMS including significant weight gain, immunosuppression, and physical inactivity. These risk factors have been shown to be partly reversible with an active lifestyle. A home-based exercise program may prove to be an effective post-transplant intervention for improving the metabolic profile of transplant recipients.

Primary objective: To evaluate the feasibility (recruitment rate, program adherence, attrition, safety, and participant satisfaction) of a 12 week individualized, virtual home-based aerobic and resistance training program in OLT and LTx recipients that are 12-18 months post-transplant. Secondary objective: To assess estimates of intervention efficacy on elements of PTMS, insulin resistance, exercise self-efficacy, and HRQL.

Hypotheses: We hypothesize that it will be feasible to recruit both OLT and LTx recipients into a home-based exercise program with ≥ 70% adherence to the prescribed exercise dose. Secondary Objective: PTMS risk factors, self-efficacy and HRQL will be improved with a home-based exercise program.

The home-based exercise group will be asked to exercise 3 to 5 times per week (≥ 150 minutes of aerobic exercises at moderate intensity) and to also complete resistance training (resistance bands or free weights) over a 12-week period with the guidance of a qualified exercise professional. The control group will be counselled by a qualified exercise professional on the importance of accumulating at least 150 minutes of moderate physical activity during the first assessment at the beginning of the study. Both groups will also receive physical activity trackers (Fitbit), exercise training or physical activity logs, and a counselling session by the dietitian at the start of the study.

A home-based exercise program may prove to be an effective post-transplant intervention for improving the metabolic profile of transplant recipients. Characterizing the feasibility, adherence, and effect estimates of home-based exercise training constitutes the first key step in promoting a healthy lifestyle in transplant recipients, and supporting the development of future trials aimed at reducing the morbidity associated with PTMS.

ELIGIBILITY:
Inclusion Criteria:

* Adult lung and liver transplant recipients 12 to 18 months post-transplant
* Presence of 2 or more metabolic risk factors (hypertension, hyperlipidemia, diabetes, obesity)

Exclusion Criteria:

* Active cardiovascular disease (recent heart attack, significant coronary artery disease on cardiac catheterization, heart failure, uncontrolled arrhythmias, chest pain, dizziness, or fainting in the last 3 months)
* Neuro-muscular disease or orthopedic limitations
* Physically active with ≥ 150 minutes/week of moderate-intensity aerobic physical activity
* Residing outside the province of Ontario

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Recruitment | When recruitment is complete (approximately 18 months after study initiation)
  We will measure recruitment-success percentage and will record reasons for non-participation.
Adherence to Exercise Training | Over a 12 week period
  Adherence to the home-based exercise program (aerobic and resistance) will be measured through an exercise diary completed by participants and reviewed through weekly communication.
Study Retention | Over a 12 week period
  Retention will be assessed by measuring attrition throughout the intervention period.
Adverse Events During Exercise Training (Safety and Tolerability) | Over a 12 week period
  Adverse events with exercise training will be assessed throughout the study period.
Participant Satisfaction with Exercise Training and Study Participation (Exercise Group) | Change over the study period assessed at weeks 2, 6, and 12
  Multiple choice and free form questionnaire assessing the participants' satisfaction with the home exercise program and study intervention.
Participant Satisfaction with Study Participation (Control Group) | 12 weeks from baseline assessment
  Multiple choice and free form questionnaire assessing participants' satisfaction with the study intervention.

SECONDARY OUTCOMES:
Total Cholesterol | Change from baseline at 12 weeks
  Participants will undergo fasting blood work to assess total cholesterol levels.
Triglycerides | Change from baseline at 12 weeks
  Participants will undergo fasting blood work to assess triglyceride levels.
High Density Lipoprotein | Change from baseline at 12 weeks
  Participants will undergo fasting blood work to assess high density lipoprotein.
Low Density Lipoprotein | Change from baseline at 12 weeks
  Participants will undergo fasting blood work to assess low density lipoprotein.
Fasting Blood Glucose Levels | Change from baseline at 12 weeks
  Fasting blood glucose levels will be ascertained from blood testing results.
Hemoglobin A1C | Change from baseline at 12 weeks
  Hemoglobin A1C results will be assessed from bloodwork, which allows assessment of the average level of blood sugar over the previous 3 months.
Insulin Resistance | Change from baseline at 12 weeks
  Insulin resistance will be captured using the Homeostatic Model Assessment of Insulin Resistance protocol (fasting insulin * fasting blood glucose).
C-peptide Levels | Change from baseline at 12 weeks
  C-peptide levels will be analyzed via blood testing in a subset of participants on exogenous insulin therapy.
C-reactive Protein Levels | Change from baseline at 12 weeks
  C-reactive protein levels will be ascertained from blood testing results.
Health Related Quality of Life assessed with the Short-Form 36 Health Survey | Change from baseline at 12 weeks
  The Short-Form 36 Health Survey (SF-36) will be used to assess general health-related quality of life. The SF-36 consists of eight scaled scores (total score ranging from 0 to 100), with lower scores representing lower health-related quality of life.
Physical Function assessed with the Short-Physical Performance Battery | Change from baseline at 12 weeks
  The Short-Physical Performance Battery will assess participants' balance, gait speed, and ability to rise from a chair 5 times.
Physical Activity Questionnaire | Change from baseline at 12 weeks
  The Physical Activity Scale for the Elderly (PASE) is a short survey created to assess physical activity levels in older adults. The PASE uses frequency, duration, and intensity level of physical activities over one week to assign a score (ranging from 0 to 793), with higher scores indicating greater levels of physical activity.
Self-Efficacy with Exercise Training (Exercise Group) | Change from baseline at 2, 6, and 12 weeks
  The Exercise Self-Efficacy Scale (ESES) is a 4-point rating Likert scale in which participants rate their confidence with carrying out their regular physical activities and exercise. The ESES uses a 100-point percentage scale, ranging from 0% (not at all confident) to 100% (highly confident). Higher scores represent higher self-efficacy to exercise.
Self-Efficacy with Exercise Training (Control Group) | Change from baseline at 12 weeks
  The Exercise Self-Efficacy Scale (ESES) is a 4-point rating Likert scale in which participants rate their confidence with carrying out their regular physical activities and exercise. The ESES uses a 100-point percentage scale, ranging from 0% (not at all confident) to 100% (highly confident). Higher scores represent higher self-efficacy to exercise.
Nutritional Questionnaire | Change from baseline at 12 weeks
  The Rapid Eating and Activity Assessment for Patients (REAP) survey assesses nutrient intake and helps with lifestyle counseling. The survey contains 27 questions with higher scores indicating higher diet quality (score range, 27 to 81).
Lifestyle and Environmental Questionnaire | Baseline
  The Lifestyle and Environmental Questionnaire is a questionnaire developed by our research team to assess familiarity and comfort levels surrounding technology, barriers to exercise and assess previous experience with exercise. It is composed of 10 multiple-choice questions with each question assessed independently.

OTHER OUTCOMES:
Liver Fibrosis | Change from baseline at 12 weeks
  A liver Fibroscan (transient elastography) assessment will be performed in a subset of liver transplant recipients to assess the degree of liver fibrosis (thickening/scarring of tissues). The fibrosis result is measured in kilopascals (kPa). This test is optional for study participants.
Fat Free Mass Index | Change from baseline at 12 weeks
  Fat-free mass index will be evaluated using bioelectrical impedance. This test is optional for study participants.
Body Fat Mass Index | Change from baseline at 12 weeks
  Body Fat Mass Index will be evaluated using bioelectrical impedance. This test is optional for study participants.
Electrocardiogram | Baseline
  12 Lead Electrocardiogram will be performed in all study participants. The following electrocardiogram parameters (p wave, QRS complex, QT interval, T waves, and ST segments) will be assessed to ensure they are within normal limits before starting exercise program.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Rozenberg, MD PhD, Principal Investigator — University Health Network /University of Toronto
Locations (1):
- University Health Network - Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rozenberg D, Santa Mina D, Nourouzpour S, Camacho Perez E, Stewart BL, Wickerson L, Tsien C, Selzner N, Shore J, Aversa M, Woo M, Holdsworth S, Prevost K, Park J, Azhie A, Huszti E, McLeod E, Dales S, Bhat M. Feasibility of a Home-Based Exercise Program for Managing Posttransplant Metabolic Syndrome in Lung and Liver Transplant Recipients: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2022 Mar 23;11(3):e35700. doi: 10.2196/35700. PMID 35319467